CLINICAL TRIAL: NCT03802240
Title: A Randomized, Double-blind, Multi-center, Phase III Clinical Study Assessing the Efficacy and Safety of Sintilimab ± IBI305 Combined With Pemetrexed and Cisplatin in Patients With EGFR-mutant Locally Advanced or Metastatic Non-squamous Non-small Cell Lung Cancer Who Have Failed Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI) Treatment (ORIENT-31)
Brief Title: Sintilimab ± IBI305 Plus Chemotherapy (Pemetrexed + Cisplatin) for EGFRm + Locally Advanced or Metastasis Non-Squamous NSCLC Patients After EGFR-TKI Treatment Failure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIBI338A301
Record Dates: First submitted 2019-01-07; First posted 2019-01-14 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — sintilimab; Pemetrexed; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sintilimab +IBI305+Pemetrexed+Cisplatin (Experimental): Drug: Sintilimab 200mg IV Q3W Other Name: IBI308
  Drug: IBI305 15mg/kg IV Q3W
  Drug: Pemetrexed 500mg/m2 IV Q3W
  Drug: Cisplatin 75mg/m2 IV Q3W
  Interventions: Drug: Sintilimab; Drug: IBI305; Drug: Pemetrexed; Drug: Cisplatin
- Sintilimab +Placebo2+Pemetrexed+Cisplatin (Experimental): Drug: Sintilimab 200mg IV Q3W Other Name: IBI308
  Drug: Pemetrexed 500mg/m2 IV Q3W
  Drug: Cisplatin 75mg/m2 IV Q3W
  Drug: Placebo2 Placebo2 IV Q3W
  Interventions: Drug: Sintilimab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Placebo2
- Placebo1+Placebo2+Pemetrexed+Cisplatin (Active Comparator): Drug: Pemetrexed 500mg/m2 IV Q3W
  Drug: Cisplatin 75mg/m2 IV Q3W
  Drug: Placebo1 Placebo1 IV Q3W
  Drug: Placebo2 Placebo2 IV Q3W
  Interventions: Drug: Pemetrexed; Drug: Cisplatin; Drug: Placebo1; Drug: Placebo2

INTERVENTIONS:
Drug: Sintilimab — 200mg IV Q3W
  Other Names: IBI308
  Arms: Sintilimab +IBI305+Pemetrexed+Cisplatin; Sintilimab +Placebo2+Pemetrexed+Cisplatin
Drug: IBI305 — 15mg/kg IV Q3W
  Arms: Sintilimab +IBI305+Pemetrexed+Cisplatin
Drug: Pemetrexed — 500mg/m2 IV Q3W
Drug: Cisplatin — 75mg/m2 IV Q3W
Drug: Placebo1 — Placebo1 IV Q3W
  Arms: Placebo1+Placebo2+Pemetrexed+Cisplatin
Drug: Placebo2 — Placebo2 IV Q3W
  Arms: Placebo1+Placebo2+Pemetrexed+Cisplatin; Sintilimab +Placebo2+Pemetrexed+Cisplatin

SUMMARY:
The anti-tumor activity of anti-PD-1 therapy and VEGF inhibitor in TKI-resistant EGFR-mutated non-squamous NSCLC Chinese patients will be investigated in this clinical trial.

ELIGIBILITY:
Main Inclusion Criteria:

1. Signed written informed consent before any trial-related processes;
2. Age ≥ 18 years and <75 years male or females;
3. Has a histologically or cytologically confirmed stage IIIB/IIIC (American Joint Committee on Cancer [AJCC] 8th edition) NSCLC that is unresectable and not fit for radical concurrent chemoradiotherapy, or metastatic / recurrent non-squamous NSCLC;
4. Patients with EGFR mutation confirmed by tumor histology or cytology or hematology prior to EGFR-TKI treatment
5. EGFR-TKI resistance, confirmed by RECIST 1.1
6. The investigator confirms at least one measurable lesion according to RECIST 1.1. A measurable lesion located in the field of previous radiation therapy or after local treatment may be selected as a target lesion if progression is confirmed; The Eastern Cancer Cooperative Group (ECOG) performance score of 0 or 1;

Exclusion criteria:

1. Squamous cell > 10%. If small cell types are present, the subject is not eligible for inclusion.;
2. Has previously received systemic anti-tumor treatment other than EGFR-TKI for or advanced non-squamous NSCLC (including cytotoxic chemotherapy for radiotherapy, do not include other systemic treatment for other cured tumors);
3. Has previously received the following therapies: anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or any other stimulatory or inhibitory agents of T cell receptors (eg CTLA-4, OX-40, CD137);
4. Has received EGFR-TKI treatment within 2 weeks;
5. Diagnosed of immunodeficiency or has received systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drugs.
6. History of pneumonitis requiring steroid therapy or the presence of interstitial lung disease within 1 year prior to the first dose of study drugs;
7. Symptomatic central nervous system metastases (CNS) metastasis and/or cancerous meningitis.

   Hemoptysis within 3 months,
8. Full-dose oral or parenteral anticoagulant or thrombolytic agent for 10 consecutive days within 2 weeks. prophylactic use of anticoagulants is allowed;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 492 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
PFS (Progression Free Survival) | Time from randomization to first documented disease progression (radiographic) assessed by Independent Imaging Assessment Committee (IRRC) or death due to any cause. up to 24month

SECONDARY OUTCOMES:
OS (Overall Survival) | Time from randomization to the death of the subject due to any cause assessed up to 36 months.
ORR (overall response rate) | The proportion of subjects who have a complete response (CR) or a partial response (PR) assessed up to 24 months.
PFS (Progression Free Survival) | Time from randomization to first documented disease progression (radiographic) assessed by investigator or death due to any cause up to 24 month.
DCR(Disease control rate ) | The proportion of subjects in the analysis population who had a complete response (CR) or partial response (PR) or stable disease (SD) up to 24 month.
TTR（Time to objective response ) | For subjects with CR or PR, defined as the time from randomization to the first documented CR or PR up to 24 month.
DOR(Duration of response) | For subjects with CR or PR, defined as the time from the first documented CR or PR to disease progression or death up to 24 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Lu S, Wu L, Jian H, Cheng Y, Wang Q, Fang J, Wang Z, Hu Y, Han L, Sun M, Miao L, Ding C, Cui J, Wang K, Li B, Li X, Ye F, Liu A, Pan Y, Cang S, Zhou H, Sun X, Shen Y, Wang S, Zhang W, He Y. Sintilimab plus chemotherapy for patients with EGFR-mutated non-squamous non-small-cell lung cancer with disease progression after EGFR tyrosine-kinase inhibitor therapy (ORIENT-31): second interim analysis from a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Respir Med. 2023 Jul;11(7):624-636. doi: 10.1016/S2213-2600(23)00135-2. Epub 2023 May 5. PMID 37156249
- [Derived] Lu S, Wu L, Jian H, Chen Y, Wang Q, Fang J, Wang Z, Hu Y, Sun M, Han L, Miao L, Ding C, Cui J, Li B, Pan Y, Li X, Ye F, Liu A, Wang K, Cang S, Zhou H, Sun X, Ferry D, Lin Y, Wang S, Zhang W, Zhang C. Sintilimab plus bevacizumab biosimilar IBI305 and chemotherapy for patients with EGFR-mutated non-squamous non-small-cell lung cancer who progressed on EGFR tyrosine-kinase inhibitor therapy (ORIENT-31): first interim results from a randomised, double-blind, multicentre, phase 3 trial. Lancet Oncol. 2022 Sep;23(9):1167-1179. doi: 10.1016/S1470-2045(22)00382-5. Epub 2022 Jul 28. PMID 35908558